CLINICAL TRIAL: NCT05610436
Title: Post-Covid Condition Monitoring Cohort: Evaluation of the Evolution of Symptomatology, Patient Profile and Associated Prognostic Factors
Brief Title: Post-Covid Condition Cohort: Evolution of Symptomatology, Patient Profile and Associated Prognostic Factors
Acronym: SYNPOCov
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GOEHRINGER François, Principal Investigator, clinical physician, Infectious Diseases department, Central Hospital, Nancy, France
Other Study IDs: 2022PI148
Record Dates: First submitted 2022-10-20; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-10

CONDITIONS: Long COVID; Post-Acute COVID-19; Post-Acute COVID19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our cohort is to collect prospectively, in a standardized and exhaustive manner, the health data of patients referred to the CAPCoV, our holistic referal post covid clinics for post-covid condition in order to be able to identify typical profiles of patients suffering from post covid syndrome and to follow the evolution of their disease over time.

ELIGIBILITY:
Inclusion Criteria:

* outpatients treated in the Nancy University Hospital Long Covid Support and Care Center for post-Covid condition according to WHO definition

Exclusion Criteria:

* patient opposing the processing for research purposes of their data collected in routine care for their care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients treated in the Nancy University Hospital Long Covid Support and Care Center for post-Covid condition according to WHO definition
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Symptoms | every 6 months up to 3 years
  Symptoms collected in a standardized manner during consultations, their persistence over time, their evolution (improvement, stagnation, worsening) and their severity (mild, moderate, severe)

SECONDARY OUTCOMES:
Medical history | baseline
fatigue | every 6 months up to 3 years
  Chalder scale: range 0 to 33, >22/33 classified severe
Dyspnea | every 6 months up to 3 years
  mMRC
Cognitive impairement | every 6 months up to 3 years
  Montréal Cognitive Assessment : range 0 to 30, <26/30 classified pathologic
inappropriate hyperventilation syndrome | every 6 months up to 3 years
  Nijmegen score: range 0 to 64, >23/34 classified "possible inapropriate hyperventilation" syndrome"
additional examinations | every 6 months up to 3 years
  Biology, imaging

CONTACTS AND LOCATIONS:
Overall Officials: Francois GOEHRINGER, MD, Principal Investigator — Infectious Diseases Department, Nancy University Hospital,F-54000 Nancy, France.
Locations (1):
- Nancy University Hospital, Vandœuvre-lès-Nancy, Grand Est, France